CLINICAL TRIAL: NCT00447499
Title: A Multi Center Open Label Study to Assess the Ability of Subjects With Acromegaly or Their Partners to Administer Somatuline Autogel
Brief Title: Assessment of the Ability of Subjects With Acromegaly or Their Partners to Administer Somatuline Autogel
Acronym: SALSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS315
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Results first posted 2010-12-20 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Acromegaly
Keywords: Acromegaly; Somatostatin Analogs; Somatuline® Autogel®; lanreotide; growth hormone; IGF-1; Inappropriate Growth Hormone Secretion Syndrome; Somatotropin Hypersecretion Syndrome; Inappropriate GH Secretion Syndrome
MeSH Terms: conditions — Acromegaly | interventions — lanreotide

ARMS (1):
- Somatuline Autogel (lanreotide acetate) (Experimental): Somatuline Autogel (lanreotide acetate) Injection
  Interventions: Drug: Somatuline Autogel (lanreotide acetate); Behavioral: Home administration

INTERVENTIONS:
Drug: Somatuline Autogel (lanreotide acetate) — Injections
Behavioral: Home administration — Questionnaire

SUMMARY:
The purpose of this study is to determine whether subjects with acromegaly (or their partners) are able to self administer Somatuline Autogel at home.

DETAILED DESCRIPTION:
Clinical experience with Somatuline Autogel to date has raised the possibility of self or partner injection. Previous microparticle somatostatin analogue formulations required careful reconstitution and as a result the cost of the analogues and the inconvenience of reconstitution meant self or partner injection was not a viable option.

Somatuline Autogel does not require reconstitution as it comes ready-mixed in a pre-filled syringe, thus making it more user-friendly than its predecessor and introducing the possibility of self or partner injection.

Patients with acromegaly often travel considerable distances every 28 days in order to receive their somatostatin analogue injections in the clinic. If Somatuline Autogel can be safely administered unsupervised, while maintaining disease control, this could offer patients considerable benefits in terms of reduced frequency of visits to the clinic.

This study is designed to allow suitably motivated patients with acromegaly or their partners to learn how to successfully inject Somatuline Autogel while maintaining their mean GH level control. Disease control in these patients will be assessed by comparing their GH and IGF-1 levels to accepted medical standards for control of acromegaly and by comparing the levels of GH and IGF-1 control achieved with baseline values.

ELIGIBILITY:
Inclusion Criteria:

* The subject must give signed informed consent before any study-related activities.
* The partner, if applicable, must give signed informed consent before administration of Somatuline Autogel.
* The subject must be able to understand the protocol requirements.
* The subject must have a clinical diagnosis of acromegaly due to pituitary tumor.
* The subject must be treated with a long-acting somatostatin analogue with or without a dopamine agonist and have been on the current medical regimen for at least 3 months prior to screening and have IGF-1 levels no higher than 10% above the upper limit of the normal range for age and gender at the screening visit or be somatostatin analogue naïve (if the subject is treated with a dopamine agonist he/she must have been on the current dose for at least 3 months prior to screening).
* Subjects who are treated with a dopamine agonist have to stay on their current dose for the duration of the study.
* Switch subjects must have had their last pre-study routine clinical treatment with Sandostatin LAR between 28 and 35 days before Visit 2 (enrollment).
* The subject must be able to store the study medication in a refrigerator in his/her own or his/her partner's home.
* The subject must be ≥18 years of age.
* Female subjects of childbearing potential must use adequate contraception.
* Female subjects of childbearing potential who are taking oral contraceptives must agree to stay on their current contraceptive dose for the duration of the study.
* The partner, if applicable, must be ≥18 years of age.

Exclusion Criteria:

* The subject has had pituitary surgery (adenomectomy) within 3 months prior to screening.
* The subject has received pituitary radiotherapy within 3 years prior to screening.
* The subject has received a GH receptor antagonist within 6 months prior to screening.
* The subject is currently on a higher dose of Sandostatin LAR than 30mg q28d
* The subject is pregnant or breastfeeding.
* The subject has clinically significant renal or hepatic abnormalities.
* The subject has a symptomatic, untreated biliary lithiasis.
* The subject has uncontrolled diabetes or thyroid disease.
* The subject has a known hypersensitivity to any of the test materials or related compounds.
* The subject is unable or unwilling to comply with the protocol.
* The subject has received any investigational drug within 30 days prior to screening.
* The subject has participated in a medical device study within 30 days prior to screening.
* The subject has previously participated in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen (formerly Tercica)
Locations (13):
- United States (13):
  - Diabetes and Endocrine Associates, La Mesa, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Denver VA Medical Center, Denver, Colorado
  - Northwestern University The Feinberg School of Medicine, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachussetts General Hospital, Boston, Massachusetts
  - NYU School of Medicine, New York, New York
  - Columbia University, New York, New York
  - Sisters of Charity Hospital, Buffalo, Williamsville, New York
  - Oregon Health and Science University, Portland, Oregon
  - Research Institute of Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Salvatori R, Nachtigall LB, Cook DM, Bonert V, Molitch ME, Blethen S, Chang S; SALSA Study Group. Effectiveness of self- or partner-administration of an extended-release aqueous-gel formulation of lanreotide in lanreotide-naive patients with acromegaly. Pituitary. 2010 Jun;13(2):115-22. doi: 10.1007/s11102-009-0207-x. PMID 19898989

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled on 6/28/2007 and last patient completed on 12/11/2008. The study enrolled patients with a diagnosis of acromegaly due to a pituitary tumor. patients were recruited from the patient populations of participating investigators and from referrals from other clinics and private practices. A competitive recruitment was used.
Pre-assignment Details: Patient had been treated with a long-acting somatostatin analog for at least 3 months prior to Screening, must have had IGF-1 levels < 10% above the upper limit of normal range, OR the patient was somatostatin analog-naïve (if the patient was treated with a dopamine agonist, he/she must have been on the dose for >= 3 months prior to Screening)
Groups:
- Somatuline Autogel (Lanreotide Acetate) Injection: Somatuline Autogel (lanreotide acetate) Deep Sub-cutaneous Injection 60 to 120 mg every 28 days
Period: Overall Study
Arm/Group | Somatuline Autogel (Lanreotide Acetate) Injection
Started | 59
Completed | 52
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Patient Decision | 4
Not completed — Sponsor Decision | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Somatuline Autogel (Lanreotide Acetate) Injection
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 47
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 59
Dopamine Agonist Treatment [Number; unit: Participants]
  Yes | 11
  No | 33
  Missing | 15
Previous Pituitary Surgery [Number; unit: participants]
  Yes | 52
  No | 7
Prior Somatostatin Analogue Treatment [Number; unit: participants]
  Yes | 38
  No | 6
  Missing | 15
Duration of Acromegaly [Mean (Standard Deviation); unit: Years] | 7.8 (6.7)
Time Since Last Pituitary Surgery [Mean (Standard Deviation); unit: Years] | 6.7 (6.2)
Time Since Last Somatostatin Analogue Treatment [Mean (Standard Deviation); unit: Days] | 78.8 (173.3)
Weight [Mean (Standard Deviation); unit: Kg] | 93.0 (23.8)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects or Their Partners That Are Competent to Self-administer Somatuline Autogel at the End of the Study, (Week 24/Early Termination), as Assessed by the Competence Questionnaire Score.
Description: The primary efficacy endpoint was the percentage of patients (Switch and other) or their partners who were competent to self-administer lanreotide at the end of the study (Week 24/Early Termination), as assessed by the Assessment of Competence Questionnaire (0 = 'No' and 1 = 'Yes').
Time Frame: 24 weeks
Population: All patients enrolled in the study. Patients either switched directly from octreotide (Switch patients, n = 33) or were somatostatin analogue treatment-naïve, or were not currently on octreotide treatment at study start (Other patients, n = 26).
Measure: Number; unit: Percentage of Participants
Arm/Group | Somatuline Autogel (Lanreotide Acetate) Injection
Number analyzed (Participants) | 54
Percentage of Participants | 98

2. Secondary Outcome: Percentage of Switch Subjects Who Find Self-administration of Somatuline Autogel Convenient as Assessed by the Subject Convenience Questionnaire Score.
Description: Experienced Convenience of Somatuline® Autogel® Injections was assessed by the subject as: Very convenient; somewhat convenient; neither convenient nor inconvenient; Neither convenient nor inconvenient; Somewhat inconvenient; very inconvenient.
Time Frame: 24 weeks
Population: Patients switched directly from octreotide.
Measure: Number; unit: Percent of Participants
Arm/Group | Somatuline Autogel (Lanreotide Acetate)/Switch Patient
Number analyzed (Participants) | 32
Percent of Participants | 91

3. Secondary Outcome: Percentage of Switch Subjects That Have IGF-1 Levels Within the Normal Range for Age and Gender at the End of the Study
Description: Blood sample was collected while subject is in a fasting state or non-fasting state for measuring the level of IGF-1.
Time Frame: 24 weeks
Population: Patients switched directly from octreotide who had IGF-1 level measured at the end of study.
Measure: Number; unit: Percent of Participants
Arm/Group | Somatuline Autogel (Lanreotide Acetate)/Switch Patient
Number analyzed (Participants) | 32
Percent of Participants | 94

4. Secondary Outcome: Percentage of Switch Subjects That Have Glucose Suppressed GH Levels ≤ 2.5 ng/ml at the End of the Study, Week 24/Termination.
Description: Blood samples taken before and 60 and 120 min after glucose load from fasting patient.
Time Frame: 24 Weeks
Population: Patients switched directly from octreotide who had GH level measured at the end of study.
Measure: Number; unit: Percent of Participants
Groups:
- Somatuline Autogel (Lanreotide Acetate): Somatuline Autogel (lanreotide acetate) Injection/Switch Patient
Arm/Group | Somatuline Autogel (Lanreotide Acetate)
Number analyzed (Participants) | 26
Percent of Participants | 89

5. Secondary Outcome: Change of GH Concentration Levels From Basaeline to Week 24 in Switch Patients
Description: Blood samples taken before and 60 and 120 min after glucose load from fasting patient.
Time Frame: 24 Weeks
Population: Patients switched directly from octreotide who had GH level measured at the end of study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Somatuline Autogel (Lanreotide Acetate) Injection
Number analyzed (Participants) | 26
ng/mL | -0.3 (1.3)

6. Secondary Outcome: Total Symptom Questionnaire Score at Week 24/Termination
Description: Acromegaly symptoms are sweating, snoring, joint pain, headache and fatigue. Each symptom was scored as -2 = 'always', -1 = 'most of the time', 0 = 'sometimes', 1 = 'rarely and 2 = 'never'. The total score was used to evaluate symptom control in each patient at Week 0 and Week 24/Termination. The total worst score is -10 and best score is 10.
Time Frame: 24 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: On a Scale from -10 to 10
Arm/Group | Somatuline Autogel (Lanreotide Acetate) Injection
Number analyzed (Participants) | 59
On a Scale from -10 to 10 | 0.9 (3.6)

7. Secondary Outcome: Total Health Care Professional Convenience Questionnaire Score at Week 24/Termination
Description: Healthcare professional convenience questionnaires are: Confident the Subject Properly Administering the Injection; Subject Complained About Pain When Administering the Injection; Subject Appreciated the Option of Self-Injection at Home. Each Healthcare professional convenience questionnaire was scored -2, -1, 0, 1 and 2; from most negative to most positive response. A total score across all questions was calculated and was used to evaluate the convenience. The worst total score is -6 and best total score is 6.
Time Frame: 24 weeks
Population: All patients enrolled in the study. Patients either switched directly from octreotide (Switch patients, n = 33) or were somatostatin analogue treatment-naïve, or were not currently on octreotide treatment at study start (Other patients, n = 26). Fifty-six of patients had data at Week 24.
Measure: Mean (Standard Deviation); unit: On a Scale from -6 to 6
Arm/Group | Somatuline Autogel (Lanreotide Acetate) Injection
Number analyzed (Participants) | 56
On a Scale from -6 to 6 | 4.6 (1.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected until 30 days after last subject visit or until resolution. Adverse event collection for an individual subject was up to 8 months. Across study adverse event reporting continued for a total of 1 years 7 months.
Arm/Group | Somatuline Autogel (Lanreotide Acetate) Injection
Serious Adverse Events (participants affected / at risk) | 5/59
Other Adverse Events (participants affected / at risk) | 52/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somatuline Autogel (Lanreotide Acetate) Injection (N=59)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Thyroid gland Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somatuline Autogel (Lanreotide Acetate) Injection (N=59)
Abdominal Pain (Gastrointestinal disorders) | 9 (17)
Abdominal Pain Upper (Gastrointestinal disorders) | 9 (11)
Constipation (Gastrointestinal disorders) | 3 (5)
Diarrhoea (Gastrointestinal disorders) | 28 (68)
Flatulence (Gastrointestinal disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 10 (13)
Stomach Discomfort (Gastrointestinal disorders) | 3 (6)
Asthenia (General disorders) | 3 (3)
Fatigue (General disorders) | 7 (14)
Injection Site Irritation (Gastrointestinal disorders) | 5 (5)
Injection Site Mass (General disorders) | 4 (6)
Injection Site Nodule (General disorders) | 3 (9)
Injection Site Pain (General disorders) | 12 (18)
Injection Site Pruritus (General disorders) | 5 (5)
Injection Site Swelling (General disorders) | 5 (7)
Influenza (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (15)
Back Pain (Musculoskeletal and connective tissue disorders) | 8 (12)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 (12)
Dizziness (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 16 (37)
Paraesthesia (Nervous system disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No